CLINICAL TRIAL: NCT05438251
Title: Exploring the Effect of Fespixon Cream for the Treatment of Diabetic Foot Ulcers (TEXAS 3A, 3B)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume.
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Collaborators: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ON101CLAS08
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Foot Ulcer (DFU)
Keywords: ON101; Fespixon; Diabetic Foot Ulcer; TEXAS 3A/3B
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Uncontrolled; Open-label; Randomized: N/A; Single Arm; Duration of treatment: up to 12 weeks; Titration: no; One-center(Taiwan)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diabetic Foot Ulcers (TEXAS 3A, 3B) (Experimental): 1. Name: Fespixon Cream
  2. Dosage form: Topical cream, 15 g ointment per tube
  3. Active ingredients: 1.25% extracts of Plectranthus amboinicus (PA-F4, 0.25%) and Centella asiatica (S1, 1%)
  4. Dose(s): Apply 1 cc per 5 cm^2 ulcer size (approximately 2 mm in thickness)
  5. Dosing schedule: Apply twice a day
  6. Duration: up to 12 weeks
  Interventions: Drug: Fespixon Cream

INTERVENTIONS:
Drug: Fespixon Cream — 1. Name: Fespixon Cream
  2. Dosage form: Topical cream, 15 g ointment per tube
  3. Active ingredients: 1.25% extracts of Plectranthus amboinicus (PA-F4, 0.25%) and Centella asiatica (S1, 1%)
  4. Dose(s): Apply 1 cc per 5 cm^2 ulcer size (approximately 2 mm in thickness)
  5. Dosing schedule: Apply twice a day
  6. Duration: up to 12 weeks
  Other Names: ON101 cream

SUMMARY:
A Research Study to evaluate the therapeutic effect of Fespixon cream in patients suffering from DFU (UTWCS Grade III-A or III-B) by measuring the change of grade of UTWCS (University of Texas Diabetic Wound Classification system), wound area reduction, infection control, and incidence of treatment-emergent adverse event (TEAE).

DETAILED DESCRIPTION:
This study is designed as a single-arm, open-label, one-center study to evaluate the therapeutic effect of Fespixon cream in patients suffering from DFU (UTWCS Grade III-A or III-B). The duration of this study is: run-in/ screening phase (7 days ± 3 days); treatment phase (12 weeks); follow-up phase (2 weeks ± 4 days), and visits are conducted every week during the run-in/ screening phase and every 2 weeks during the treatment phase and follow-up phase for a total of 9 visits. During the treatment phase, the Fespixon cream will be applied to the target ulcer twice a day for a maximum period of 12 weeks, until the target ulcer downgrade from UTWCS grade III-A or III-B to I-A, I-B, II-A, or II-B for two consecutive visits at least 2 weeks apart, or until the subject exited the study as treatment failure. After that, all subjects regardless of wound grade-down at the end of the treatment phase will be followed for 2 weeks. During the follow-up phase, standard of care or other treatment modalities (with an exception of investigational treatment/ medications) will be used for all subjects at the discretion of the investigator.

At each visit, the size and changes of the target ulcer are recorded by photographing. The target ulcer area in the photo is calculated using Image-Pro® Plus software.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, male or female, aged 20 to 80 years (inclusive) with Type 1 or Type 2 diabetes undergoing therapy for glycemic control using available diabetes drugs including insulin.
2. Subject has a glycosylated hemoglobin, HbA1c ≤ 12%.
3. Presence of at least one diabetic foot ulcer that meets all of the following criteria:

   1. A full-thickness ulcer of UTWCS Grade III-A or III-B
   2. Ulcer size (area) is >2 cm^2 and ≤30 cm^2 (post-debridement at time of enrollment)
   3. Ulcer is located on or below the malleoli.
   4. Ulcer presents for >1 week (at time of enrollment).
   5. There is a minimum 3 cm margin between the qualifying Target Ulcer and any other ulcers on the specified foot, (post-debridement).
   6. The infection severity of the target ulcer is defined as uninfected, mild, or moderate infection by IDSA/ IWGDF Guidelines. (IDSA/IWGDF-defined severe infection would be excluded)

   Note:
   * If the subject has more than one qualifying diabetic foot ulcer, the most severe ulcer will be designated as the target ulcer; meanwhile, the depth of the wound will the consideration prior to the area of the wound.
   * Any foot infection with the following signs of a systemic inflammatory response syndrome is defined as severe infection according to IDSA Infection Severity. This response is manifested by two or more of the following conditions:

     1. temperature>38℃ or <36℃
     2. heart rate > 90 beats/minute
     3. respiratory rate > 20 breaths/minute or PaCO2 < 32 mmHg
     4. WBC ( white blood cell count ) < 4.0 X 10^9 cells/ L； > 12.0 X 10^9 cells/ L or ≥ 10% immature (band) forms.
4. Subject has adequate vascular perfusion of the affected limb, confirmed by Ankle-Brachial Index (ABI) ≥ 0.8 and < 1.3, or transcutaneous pressure of oxygen (TcPO2) ≥ 30 mmHg on at least one lead to ensure no serious embolisms / no serious clogging of blood vessels.
5. Subject, if female of child-bearing potential, have a negative serum/urine pregnancy test at screening, must not be breastfeeding, and willing to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectable, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and/or who have been sterilized).
6. Subject is willing to use an off-loading device for the target ulcer on the plantar while ambulation for the duration of the study; the study institution will provide the off-loading devices.
7. Subject / identified caregiver trained on the study procedures is able and willing to comply with study procedures.
8. A signed and dated informed consent form has been obtained from the subject prior to any study-related procedures being performed.

Exclusion Criteria:

1. Other laboratory values at Screening of:

   1. Liver function studies [Total bilirubin, aspartate aminotransferase (AST), and alanine transaminase (ALT)] > 3x the upper limit of normal
   2. Albumin < 2.5 g/dL
2. Presence of any clinically significant medical condition(s) in medical history during the screening period that, in the opinion of the investigator, could interfere with wound healing, including but not limited to the following:

   1. Acute or unstable Charcot foot
   2. Current sepsis
   3. Active malignant disease. A subject, who has had a malignant disease in the past, was treated, and is currently disease-free, may be considered for study entry
   4. Acquired immune deficiency syndrome (AIDS) or HIV positive
3. Has a known hypersensitivity to any of the investigational drug or the related components
4. X-ray or MRI scan is as a mandatory screening to rule out osteomyelitis
5. Subject is currently receiving (i.e., within 30 days of enrollment visit) or scheduled to receive any of the following medication or therapies, which could interfere with wound healing during the course of the study.

   1. immunosuppressant (including chronic systemic corticosteroids)
   2. cytotoxic chemotherapy
   3. cytostatic therapy
   4. autoimmune disease therapy
   5. lower limb revascularization surgery (e.g., angioplasty, artery bypass surgery)
   6. growth factors
   7. hyperbaric oxygen therapy
   8. bioengineered tissue or skin substitutes (ADM)
   9. application of topical steroids to the ulcer
   10. use of any investigational drug(s)
6. A psychiatric condition (e.g., suicidal ideation), current or chronic alcohol or drug abuse, determined from the subject's medical history, which, in the opinion of the investigator, may pose a threat to subject compliance.
7. Subjects who need to stand continuously for more than 4 hours/day and have difficulty complying with off-loading instructions.
8. Has any other factor which may, in the opinion of the investigator, compromise participation and/or follow-up in the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Incidence of the grade down of the target ulcer | 12 weeks
  Ulcer grade down is defined as ulcer downgrading from 3A or 3B to 1A, 1B, 2A, or 2B confirmed at two consecutive study visits 2 weeks apart.
Time to the ulcer grade down | 12 weeks
  * Ulcer grade down is defined as ulcer downgrading from 3A or 3B to 1A, 1B, 2A, or 2B confirmed at two consecutive study visits 2 weeks apart.
  * Time to the ulcer grade down was defined as "time to the first visit of ulcer grade down of the target ulcer."

SECONDARY OUTCOMES:
Mean change from baseline in the target ulcer area confirmed by Image-Pro® Plus calculation of the wound area | 12 weeks
  The target ulcer area at each visit is confirmed by Image-Pro® Plus software and presented as a mean change from the baseline.
Percentage change from baseline in the target ulcer area confirmed by Image-Pro® Plus calculation of the wound area | 12 weeks
  The target ulcer area at each visit is confirmed by Image-Pro® Plus software and presented as a percentage change from the baseline.
Percentage of ulcer improvement | 12 weeks
  Ulcer improvement is defined as ulcer downgrading from 3A or 3B to 1A, 1B, 2A, or 2B confirmed at two consecutive study visits 2 weeks apart.

CONTACTS AND LOCATIONS:
Overall Officials: Shyi-Gen Chen, VP, Study Director — Oneness Biotech Co., Ltd.
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No